CLINICAL TRIAL: NCT03719066
Title: Effect of Extended Dose Intervals on the Immune Response to Oral Cholera Vaccine in Cameroon
Brief Title: Extended Dose Intervals With Oral Cholera Vaccine in Cameroon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Meilleur Accès aux Soins de Santé (M.A. Santé) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8114
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Adverse Reaction to Cholera Vaccine; Cholera Vaccination Reaction
Keywords: cholera; oral cholera vaccine; vibriocidal titer; ELISA antibodies; Adverse event following immunization
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive two doses of Shanchol oral cholera vaccine with dose intervals of either 2 weeks, 6 months or 11 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DIG 1 (dose interval group) (Active Comparator): This group will receive two doses of killed whole cell oral cholera vaccine. The second dose being administered two weeks after the first dose.
  Interventions: Biological: killed whole cell oral cholera vaccine
- DIG 2 (dose interval group) (Experimental): This group will receive two doses of killed whole cell oral cholera vaccine. The second dose being administered 6 months after the first dose.
  Interventions: Biological: killed whole cell oral cholera vaccine
- DIG 3 (dose interval group) (Experimental): This group will receive two doses of killed whole cell oral cholera vaccine. The second dose being administered 11 months after the first dose.
  Interventions: Biological: killed whole cell oral cholera vaccine

INTERVENTIONS:
Biological: killed whole cell oral cholera vaccine — two week interval
  Other Names: Shanchol

SUMMARY:
The primary aim of this project is to determine changes in the vibriocidal geometric mean titers (GMT) in subjects who receive the second dose of oral cholera vaccine (OCV) at different intervals: 2 weeks, 6 months, or 11 months following the first dose of vaccine. Secondary aims include a) vibriocidal antibody response rates in subjects who receive OCV at 2 weeks, 6 months, or 11 months following the first dose of vaccine, b) age specific serum vibriocidal GMTs following the second dose among participants given the second dose of OCV at intervals of 2 weeks, 6 months, or 11 months following the first dose of vaccine, c) GMT and antibody response rates of Immunoglobulin A (IgA) and Immunoglobulin G (IgG) anti-lipopolysaccharide (LPS) as measured by ELISA following the second dose among participants given the second dose of OCV at intervals of 2 weeks, 6 months, or 11 months following the first dose of vaccine. The hypothesis is that the vibriocidal GMT following the second dose, when given after 6 or 12 months will not be inferior to the response when the second dose is given according to the standard interval of two weeks.

DETAILED DESCRIPTION:
This is an open label, randomized, phase 2 clinical trial of the immunogenicity of killed oral cholera vaccine (OCV) when the vaccine is administered to participants of three age cohorts (1-4 years, 5-14 years, and >14 years) and in three dose interval groups (DIGs). The subjects in each age cohort will be randomized to a DIG of 2 weeks (DIG-1), 6 months (DIG-2) or 11 months (DIG-3). A total of 180 subjects from Douala, Cameroon will be enrolled and these are equally divided between the different groups (20 per age/dose interval group). The OCV to be used in the trial is Shanchol.

Blood samples will be collected before the first dose and at intervals following the first dose depending on the dosing interval group assigned. The serum (or plasma) will be tested for antibodies to cholera.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥1 year, stratified into different age groups
2. Living in the Soboum Health Area or adjoining area
3. Good health condition, without clinically significant medical history (by participant or guardian, in case of minor)
4. Not pregnant for female subjects.
5. Available to participate for the study duration, including all planned follow-up visits for up to 18 months from screening.
6. Signed informed consent -

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition (Examples include: Diagnosis and treatment of tuberculosis (TB) or HIV; renal insufficiency; hepatic disease; oral or parenteral medication known to affect the immune function , such as corticosteroids, other immunosuppressant drugs; or behavioural or memory issues)
2. Ever having received oral cholera vaccine.
3. Receipt of an investigational product (within 30 days before vaccination).
4. History of diarrhoea in 7 days prior to first dose of vaccine (defined as ≥3 unformed loose stools in 24 hours).
5. History of chronic diarrhea (lasting for more than 2 weeks in the past 6 months)
6. Current use of laxatives, antacids, or other agents to lower stomach acidity?
7. Planning to become pregnant in the next 2 years

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Vibriocidal titer | two weeks after the second dose
  Geometric Mean titre of the vibriocidal titre

SECONDARY OUTCOMES:
ELISA titres | two weeks after the second dose
  IgG and IgA geometric mean titres against V cholerae LPS

CONTACTS AND LOCATIONS:
Overall Officials: David Sack, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- M.A. Sante, Douala, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
We will publish the results of this study in a peer reviewed publication and will make the data available on request after the paper has been published.
Supporting Information: CSR
Time Frame: When the manuscript is published.
Access Criteria: Researchers will need to submit a request to the investigators detailing their plans for analysis.